CLINICAL TRIAL: NCT01305018
Title: Effects of Leucine and Branched-chain Amino Acids (BCAA) Supplementation on Resistance Exercise-induced Muscle Damage and Inflammation: a Randomized, Double-blind, and Placebo-controlled Study
Brief Title: Branched-chain Amino Acids Supplementation and Resistance Exercise-induced Muscle Damage and Inflammation
Status: Suspended | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Claudia Ribeiro da Luz, University of São Paulo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 071287
Record Dates: First submitted 2011-02-25; First posted 2011-02-28 (Estimated); Last update posted 2011-05-05 (Estimated); Status verified 2011-04

CONDITIONS: Muscle Damage; Inflammation
Keywords: Branched-chain amino acids; Leucine; Muscle damage; Inflammation; supplementation; resistance exercise-induced
MeSH Terms: conditions — Inflammation | interventions — Leucine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Exercise and BCAA (Experimental)
  Interventions: Dietary Supplement: BCAA
- Exercise and Leucine (Experimental)
  Interventions: Dietary Supplement: Leucine
- Exercise and Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: BCAA — 7 g of leucine + 3,5 g of isoleucine + 3,5 g of valine per day during 9 days
  Arms: Exercise and BCAA
Dietary Supplement: Leucine — 7 g of leucine + 7 g of alanine per day during 9 days
  Arms: Exercise and Leucine
Dietary Supplement: Placebo — 14 g of alanine per day during 9 days
  Arms: Exercise and Placebo

SUMMARY:
This study aims to evaluate the effects of branched-chain amino acids (BCAA) supplementation on resistance exercise-induced muscle damage and inflammation.

ELIGIBILITY:
Inclusion Criteria:

* Sedentary;
* No muscle disorders;
* Must be able to swallow tablets

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2011-08; Primary Completion 2012-01 (Estimated); Study Completion 2012-08 (Estimated)

PRIMARY OUTCOMES:
Muscle maximal strength | 4 days
Muscle edema | 4 days
Muscle soreness | 4 days

SECONDARY OUTCOMES:
Muscle inflammation | 4 days
  Immunohistochemistry, protein expression.
Muscle damage | 4 days
  Serum creatine kinase

CONTACTS AND LOCATIONS:
Locations (1):
- University of São Paulo - School of Physical Education and Sports, São Paulo, São Paulo, Brazil